CLINICAL TRIAL: NCT04431895
Title: A Prospective,Single-center,Single-Arm,Single-Blind Pilot Study To Investigate The Efficacy Of Tofacitinib In Patients With Refractory Myasthenia Gravis
Brief Title: Safety And Efficacy Of Tofacitinib In Patients With Refractory Myasthenia Gravis: A Pilot Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Chongbo Zhao, Professor, Huashan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2020-019
Record Dates: First submitted 2020-06-12; First posted 2020-06-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2022-09

CONDITIONS: Myasthenia Gravis, Generalized
Keywords: myasthenia gravis; tofacitinib
MeSH Terms: conditions — Myasthenia Gravis | interventions — tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- tofacitinib 5mg twice a day (Experimental)
  Interventions: Drug: Tofacitinib 5 MG

INTERVENTIONS:
Drug: Tofacitinib 5 MG — tofacitinib 5 mg tablet administered twice a day for 6 months

SUMMARY:
This is a 6 month study that will evaluate the efficacy of 5mg tofacitinib tablet taken twice a day in patients with refractory myasthenia gravis. Twenty adult participants will receive a four month treatment of tofacitinib followed by elution for one month.

ELIGIBILITY:
Inclusion Criteria:

* fluctuating muscle weakness and fatigability classified as the Myasthenia Gravis Foundation of America (MGFA) clinical classification Type IIa-IVa;
* more than 10% amplitude decrement in low frequency repetitive nerve stimulation, and less than 10% amplitude increment in high frequency repetitive nerve stimulation;
* understanding and assigning the informed consent form, and having a good compliance with treatment.

meet all of the criteria in above as well as at least one of the below:

* refractory: insufficient response to full dose- and course- steroids treatment (0.75-1mg per kg per day for at least 3-6 months), failure to respond adequately to tacrolimus (no less than 3mg per day) for 3 months;
* severe or intolerable adverse effects from conventional immunosuppressive therapy.

Exclusion Criteria:

* positive for muscle-specific kinase (MuSK) antibodies;
* a tumor history except for thymoma;
* a history of Type B and Type C hepatitis;
* a history of tuberculosis or T-SPOT.TB tset positivity;
* hepatic, renal and cardial insufficiency (baseline: ALT/AST>50U/L;BNP>200pg/ml）;
* severe allergy or infection, or chronic or recurrent infection;
* pregnancy;
* hyperlipidemia;
* participating other clinical trials

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-06-11 (Actual); Primary Completion 2024-03-21 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Quantitative Myasthenia Gravis (QMG) Scores at Month 6 | Baseline, Month 6
  A quantitative MG scoring system (QMG Score) is essential in the objective evaluation of therapy for MG.This scoring system is based on quantitative testing of sentinel muscle groups. Total QMG score range from 0 (extreme disease severity) to 39 (none), higher score indicated less disease severity.

SECONDARY OUTCOMES:
Change From Baseline in Myasthenia Gravis-related Activities of Daily Living (MG-ADL) Scores at Month 6 | Baseline, Month 6
  The myasthenia gravis activities of daily living (MG-ADL) profile is an eight-item patient-reported scale developed to assess MG symptoms and their effects on daily activities.Total MG-ADL score range from 0 (none) to 24 (extreme disease conditions), higher score indicated more disease severity.
Change From Baseline in Myasthenia Gravis Composite (MGC) Scores at Month 6 | Baseline, Month 6
  The MGC score consists of test items that measure symptoms and signs of MG, with weighted response options. Total MGC score range from 0 (none) to 50 (extreme muscle weakness), higher score indicated more disease severity.
Change From Baseline in Myasthenia Gravis-Quality of Life Questionnaire-15 item (MG-QOL15) Scores at Month 6 | Baseline, Month 6
  The MG-QOL15 is helpful in informing the clinician about the patient's perception of the extent of and dissatisfaction with MG-related dysfunction. Total MG-QOL15 score range from 0 (none) to 60 (extreme disease severity), higher score indicated more disease severity.
Change From Baseline in Doses of Steroids at Month 6 | Baseline, Month 6
  Steroids is recommended as the first-line treatment for myasthenia gravis. Here we followed the combined doseage of steroids while administrating tofacitinib for enrolled participants.

OTHER OUTCOMES:
Change From Baseline in Serum Titers of anti-acetylcholine receptor antibodies at Week 16 | Baseline, Week 16
  Anti-acetylcholine receptor antibodies are the major pathological autoantibodies of MG. For anti-AChR antibodies-positive candidates, we followed the antibodies titers at Week 16.
Change From Baseline in Inflammatory Cytokines at Week 12 | Baseline, Week 12
  MG is an autoimmune disease manifested by impairment at the neuromuscular junction featured by weakness and fatigability. We compared the inflammatory cytokines (IL-6, IL-10, IL-17A, and IL-23) at Baseline and Week 12

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) are not available to other researchers.